CLINICAL TRIAL: NCT01096745
Title: Randomized Phase II Trial of Gemcitabine/Cisplatin Versus S-1/Cisplatin in Advanced Biliary Cancer Patients
Brief Title: Randomized Trial of Gemcitabine/Cisplatin Versus S-1/Cisplatin in Advanced Biliary Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Planning for randomized phase III trial for this issue.
Sponsor: Gyeongsang National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Dong-A University (Other); Chung-Ang University (Other)
Responsible Party: Jung Hun Kang/Assisstant Professor, Gyeongsang National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GNUHIRB-2010-5
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Biliary Tract Cancer; Locally Advanced Biliary Tract Cancer
Keywords: Gemcitabine; Cisplatin; S-1; bile duct cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Bile Duct Neoplasms | interventions — Gemcitabine; Cisplatin; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine/Cisplatin (Experimental)
  Interventions: Drug: Gemcitabine, Cisplatin
- S-1/Cisplatin (Experimental): D1-14 S-1 40mg/m2 po bid D1,D8 Cisplatin 25/m2 + N/S 150cc miv over 60mins Repeated every 3 weeks
  Interventions: Drug: S-1, Cisplatin

INTERVENTIONS:
Drug: Gemcitabine, Cisplatin — D1,D8 Gemcitabine 1000mg/m2 + N/S 150cc miv over 30mins D1,D8 Cisplatin 25/m2 + N/S 150cc miv over 60mins repeated every 3weeks
  Other Names: Gemcitabine - Gemcitane; Cisplatin - Cispulan
  Arms: Gemcitabine/Cisplatin
Drug: S-1, Cisplatin — D1-14 S-1 40mg/m2 po bid D1,D8 Cisplatin 25/m2 + N/S 150cc miv over 60mins Repeated every 3 weeks
  Other Names: S-1; TS-1; Cisplatin ; Cispulan
  Arms: S-1/Cisplatin

SUMMARY:
The purpose of this study is to compare the efficacy between gemcitabine/cisplatin and S-1/cisplatin in the first-line treatment in advanced biliary tract cancer.

DETAILED DESCRIPTION:
Standard chemotherapy regimen for biliary tract cancer(BTC) has not been established due to the difficulty associated with performing clinical trials in this field.

Gemcitabine or fluoropyrimidines, including 5-fluorouracil and S-1, are routinely used for BTC chemotherapy. The European Society for Medical Oncology (ESMO) and the National Comprehensive Cancer Network guidelines published in 2009 recommend either gemcitabine-based or fluoropyrimidine-based chemotherapy or clinical trials for first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age : older than 20
* Eastern Cooperative Oncology Group (ECOG) performance status 0 -2
* Histologically confirmed adenocarcinoma of the biliary tract
* Metastatic or unresectable biliary cancer
* No prior chemotherapy for biliary cancer
* A patient with at least one measurable primary lesion of which the diameter is confirmed to be 10mm in Spiral CT or multidetector CT (MD CT)
* Adequate bone marrow, liver, renal function

Exclusion Criteria:

* A patient with no measurable disease
* A patient who received previous palliative chemotherapy for biliary cancer
* A patient who received adjuvant chemotherapy for biliary cancer within 1year
* A patient with previous active or passive immunotherapy.
* A pregnant or lactating patient

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Time to progression | From the assigned day to the disease progression or the last day of follow-up without progression. Clinically assessment would be done every cycle (month) and radiologically assessed every 6 weeks with CT scan

SECONDARY OUTCOMES:
Response rate Overall survival Safety profile | Overall survival is measured from the first day of assignment until death or the last day of the follow-up.Clinically assessment would be done every cycle (month) and radiologically assessed every 2 cycles (6 weeks) with CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Chan Kwon, M.D., Principal Investigator — Dong-A University Hospital; Jung Hun Kang, M.D., Study Director — Gyeongsang University Hospital
Locations (1):
- Gyeongsang University Hospital, Jinju, Gyeongsangnam-do, South Korea